CLINICAL TRIAL: NCT01355198
Title: Role of HIV on Glutathione Synthesis and Oxidative Stress
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rajagopal Sekhar, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV and glutathione
Record Dates: First submitted 2011-03-30; First posted 2011-05-18 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infection; Erythrocyte Glutathione Deficiency
MeSH Terms: conditions — HIV Infections | interventions — Cysteine; Glycine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cysteine/glycine (Experimental): Subjects will be studied before and after receiving oral cysteine (as n-acetylcysteine) and glycine for 2 weeks
  Interventions: Dietary Supplement: Cysteine (as n-acetylcysteine) and glycine; Dietary Supplement: Cysteine/glycine

INTERVENTIONS:
Dietary Supplement: Cysteine (as n-acetylcysteine) and glycine — Cysteine and glycine will be supplemented at doses of 0.81 mmol/kg/d and 1.31 mmol/kg/d for 2 weeks each
Dietary Supplement: Cysteine/glycine — Subjects will receive oral dietary amino-acids (cystiene as n-acetylcysteine, and glycine)

SUMMARY:
HIV infection is associated the development of increased oxidative stress and deficiency of glutathione (GSH), the dominant endogenous antioxidant protein, but the underlying mechanisms contributing to GSH deficiency are hitherto unknown. Furthermore GSH metabolism has not been studied in HIV patients, in whom the burden of risk factors promoting oxidative stress is highest. Our previous studies in non-HIV human subjects with diabetes-related oxidative stress and GSH deficiency have demonstrated that the latter is due to decreased synthesis of GSH. Importantly, short-term dietary supplementation with the simple GSH precursor amino-acids cysteine and glycine, boosted GSH synthesis and cellular concentrations, corrected GSH deficiency, and reduced oxidative stress and oxidant damage. The current proposal will study whether (1) defective synthesis underlies GSH deficiency in patients with HIV, and will test a simple, inexpensive and rational therapy based on protein supplementation to improve GSH synthesis and concentrations and lower markers of oxidative stress and oxidant damage in these patients; (2) study if correction of GSH deficiency is asssociated with any changes in (a) impaired mitochondrial fuel oxidation in the fasted and insulin stimulated states; (b) insulin sensitivity; (c) body composition and anthropometry; (d) forearm muscle strength; (e) plasma biochemistry, and (f) quality of life indices in these subjects.

ELIGIBILITY:
Inclusion Criteria:

(1) HIV infected patients with GSH deficiency

Exclusion Criteria:

1. renal impairment (serum Creatinine above 1.5mg/dL), liver impairment (ALT and AST > 2x upper limit of normal)
2. any hormonal disorders such as hypothyroidism, hypercortisolemia, hypogonadism, or diabetes mellitus on pharmacotherapy
3. evidence of infections other than HIV in the preceding 3 months
4. subjects with plasma triglyceride concentrations of ≥ 500mg/dL on triglyceride lowering therapy
5. BMI < 20
6. established heart disease
7. Co-existing viral hepatitis B and C

Ages: 21 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Glutathione synthesis rates and concentrations | 9 hours
  Fractional and absolute synthesis rates of glutathione and its concentrations

SECONDARY OUTCOMES:
Mitochondrial fuel oxidation | Twice over 9 hours of the study on 2 occassions
  Lipolysis, fuel oxidation, and a hyperinsulinemic euglycemic clamp.
Rates of fuel kinetics | 3 hours
  Measure rate of lipolysis (from infused 13C-palmitate) and recovery of 13CO2 (from infused acetate tracer)
Insulin sensitivity | 3 hours
  Measure insulin sensitivity using a hyperglycemic euglycemic clamp
Muscle strength | Done once in each 9-hour study
Quality of life by SF36 questionnaire | Before and after

CONTACTS AND LOCATIONS:
Overall Officials: R V Sekhar, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor GCRC, Houston, Texas, United States